CLINICAL TRIAL: NCT03745950
Title: Multicenter Double Blind Randomized Phase II Trial of Olaparib vs Placebo as Maintenance Therapy in Platinum-sensitive Advanced Endometrial Carcinoma
Brief Title: UTOLA: UTerin OLAparib
Acronym: UTOLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GINECO-EN-104b
Record Dates: First submitted 2018-10-31; First posted 2018-11-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Carcinoma
Keywords: Maintenance therapy; Olaparib; Randomized, double blinded; P53 and MMR Immunohistochemistry; Phase II; progression-free survival
MeSH Terms: conditions — Endometrial Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: Olaparib vs placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olaparib (Experimental): The Olaparib arm :
  Patients will be administrated the randomized study treatment tablets orally at a dose of 300 mg twice daily until objective radiological disease progression as per RECIST (Response evaluation criteria in solid tumors) as assessed by the investigator, or unacceptable toxicity
  Interventions: Drug: Olaparib Oral Capsule
- Placebo (Placebo Comparator): The placebo arm :
  Patients will be administrated the randomized study treatment tablets orally at a dose of 300 mg twice daily until objective radiological disease progression as per RECIST as assessed by the investigator, or unacceptable toxicity
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Olaparib Oral Capsule — - Olaparib will be administrated by oral at dose of 300 mg twice daily during the induction period and in maintenance
  Arms: Olaparib
Drug: Placebo oral capsule — - Placebo will be administrated by oral at dose of 300 mg twice daily during the induction period and in maintenance
  Arms: Placebo

SUMMARY:
This is a phase IIB, national, randomized, double-blinded, comparative, multi-center study, to assess the efficacy of Olaparib as maintenance after a platinum based chemotherapy in patients with Advanced or metastatic endometrial cancer

DETAILED DESCRIPTION:
Approximately 147 patients will be randomized using an Interactive Voice Response System / Interactive web system (IVR/IWR system) in a 2:1 ratio to the treatments as specified below :

* Olaparib tablets per os 300 mg twice daily,
* Placebo tablets per os 300 mg twice daily.

Before randomization to the study :

* Patient should be without evidence of disease (NED), or in clinical complete response or in partial response or stable.
* Patient must have completed a minimum of 4 cycles of first line platinum based chemotherapy (recommended chemotherapy is carboplatine AUC 5 plus paclitaxel 175 mg/m2).

Patient will be stratified according to :

* P53 and MMR Immunohistochemistry, (Y/N)
* Response to previous chemotherapy line (Objective response versus Stable)

Patients will receive Olaparib/Placebo up to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Female Patient ≥18 years at the day of consenting to the study
* Provision of informed consent prior to any study specific procedures
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Patient with advanced/metastatic endometrial cancer not candidate to a curative treatment with surgery or radiotherapy
* Patients who have completed prior to randomization one Platine based chemotherapy for advanced disease after 6 cycles of chemotherapy (at least 4 cycles of platine). Patients must have a measurable disease according RECIST 1-1 at the initiation of the chemotherapy (cf. appendix 3)
* Patients must be prior to randomization without evidence of disease (NED) or in complete response (CR) or partial response (PR) or stable disease from the chemotherapy
* Patient should have been tested biolology for IHC : P53 and MMR within two weeks before the randomisation and (NGS; BRCA/HRD) within 3 months after the randomisation
* Patients could have been previously treated with Hormone-therapy
* Adjuvant chemotherapy or local radio-chemotherapy is allowed (with a delay of at least of 12 months). First recurrence at least 12 months after a loco-regional treatment.
* Patients pay have received external beam +/- vaginal brachytherapy
* All histologic and molecular subtypes of endometrial carcinoma will be included (including mixte histology), except carcinosarcoma, neuro-endocrine and small cells carcinoma.
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  1. Haemoglobin ≥10.0 g/dL with no blood transfusion in the past 28 days
  2. Absolute neutrophil count (ANC) ≥1.5 x 109/L
  3. Platelet count ≥100 x 109/L
  4. Total bilirubin ≤1.5 x institutional upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤5x ULN
  6. Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:
* Recovery from all reversible adverse events of previous anti-cancer therapies to baseline or CTCAE G 1, except for alopecia (any grade) and ≤ G 2 sensory peripheral neuropathy
* Able to swallow and retain oral drug
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential prior to the first dose of study treatment. (negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as: Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments/Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50/radiation-induced oophorectomy with last menses >1 year ago/chemotherapy-induced menopause with >1 year interval since last menses/surgical sterilisation (bilateral oophorectomy or hysterectomy)"
* Life expectancy > 16 weeks
* Patients is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* As this study will include patients in France, a subject will be eligible for randomization in this study only if either affiliated to, or a beneficiary of, a social security category.

For inclusion in ancillary studies If a patient declines to participate in the optional Biomarker/pharmacogenetic research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.

Exclusion Criteria:

* Patients with carcinosarcoma, neuro-endocrine and small cells histologies
* Patients who have previously received more than 1 line of chemotherapy for advanced/metastatic endometrial cancer
* Patients with a localized advanced disease that could be treated by surgery
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS)
* Patients with myelodysplastic syndrome/acute myeloid leukemia history or with features suggestive of MDS/AML.
* Patients receiving radiotherapy within 6 weeks prior to study treatment.
* Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Any previous treatment with PARP inhibitor, including olaparib.
* Clinically significant (e.g. active) cardiovascular disease, uncontrolled high blood pressure
* Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub- Arachnoids Hemorrhage (SAH) within 6 months prior to randomization.
* History or evidence of hemorrhagic disorders within 6 months prior to randomization
* Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Persistent toxicities (Common Terminology Criteria for Adverse Event (CTCAE) > grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Pregnant or lactating woman
* Participation in another clinical study with an investigational product during he chemotherapy course immediately prior to randomization.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Efficacy: Progression free survival (PFS1) according to modified Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) of Olaparib maintenance after a platinum based chemotherapy in patients with advanced or metastatic endometrial cancer | An average of 36 months

SECONDARY OUTCOMES:
To determine time from randomization until death from any cause | To be assessed around 73 months
To determine time from randomization to efficacy by progression free survival | To be assessed around 36 months
To determine time from response rate according to IHC P53, MMR, NGS BRCA/HRD, MSI | To be assessed around 36 months
To determine the overall response rate ORR | To be assessed around 30 months
To determine time from randomization to first and second subsequent therapy (TFST, TSST) | To be assessed around 36 months
To determine time from randomization until 2nd disease progression or death (PFS2) | To be assessed around 73 months
To assess the safety of Olaparib maintenance compared to placebo - Graded according to CTCAE version 4.03. | To be assessed around 36 months
  Graded according to CTCAE version 4.03. These will be collected by all patients.
To assess the tolerability of Olaparib maintenance compared to placebo - Graded according to CTCAE version 4.03. | To be assessed around 36 months
  Graded according to CTCAE (Common Terminology Criteria for Adverse Events) version 4.03. These will be collected by all patients.
To assess the effects of Olaparib on health-related quality of life (HRQoL) as measure by determining time to deterioration in Quality of life, based on EORTC QLQ-C30 (Quality Of Life Questionnaire-core 30) | to be assessed 36 months
  Health related quality of life of the patient. For all scales a high score is equivalent to worse or more problems. Range is the difference between the maximum and minimum possible value of the raw score. All items are scored from1 to 4, giving a range=3. For each scale, calculate the raw score by the addition of item responses divided by the number of items. Then a linear transformation is used to standardise the raw score, so that scores range from 0 to 100. Score= (raw score-1)/rangex100
To assess the effects of Olaparib on health-related quality of life (HRQoL) as measure by determining time to deterioration in Quality of life, based EORTC QLQ-EN24 (Quality of Life Questionnaire - Endometrial Cancer Module) | to be assessed 36 months
  To assess disease and treatment specific aspects of the quality of life of patients with endometrial cancer. A high score for the functional scales represents a high level of functioning, while a high score for the symptom scales represents a high level of symptoms or problems. Symptoms related to sexual/vaginal problems (EMSXV including item 51-53) are optional.
To assess the effects of Olaparib on health-related quality of life (HRQoL) as measure by determining time to deterioration in Quality of life, based on EORTC FA12 (Quality of life Module Measuring Cancer Related Fatigue) | to be assessed 36 months
  To assess physical, cognitive and emotional aspects of cancer-related fatigue.The higher the score, the better the QOL
To assess the effects of Olaparib on health-related quality of life (HRQoL) as measure by determining time to deterioration in Quality of life, based on Quality of Life Questionnaire EQ5D (consists of a descriptive system and the EQ VAS) | to be assessed 36 months
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
To determine efficacy by progression free survival | To be assessed around 73 months
  PFS1 is defined as the time from randomization until the date of the first objective radiological disease progression according to investigator assessment
To determine response rate according to response to the initial chemotherapy | To be assessed around 73 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, Principal Investigator — GINECO - Centre François Baclesse
Locations (36):
- France (36):
  - ICO Paul Papin, Angers
  - Institut du cancer Avignon-Provence, Avignon
  - CHRU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Chu Dijon, Dijon
  - Centre Georges François Leclerc, Dijon
  - Institut Daniel Hollard - GHM de Grenoble, Grenoble
  - Institut inter-régionaL de Cancérologie - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Saint-Joseph, Marseille
  - Centre Hospitalier de Mont-De-Marsan, Mont-de-Marsan
  - ICM Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent SAS, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancérologie du Gard - CHU de Nîmes, Nîmes
  - CHR d'Orléans, Orléans
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Hôpital Cochin, Paris
  - Institut Curie - Hopital Claudius Régaud, Paris
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Centre Henri Becquerel, Rouen
  - ICO Centre René Gauducheau, Saint-Herblain
  - CHU Saint Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Claudius Régaud, Toulouse
  - Institut de Cancérologie de Lorraine - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif